CLINICAL TRIAL: NCT02440997
Title: A Preliminary Investigation of the Efficacy of Aromatherapy in Reducing Discomfort in Youth With Chronic Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB # 15010015
Record Dates: First submitted 2015-04-22; First posted 2015-05-12 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Chronic Headache; Migraine Headache; Headache
Keywords: aromatherapy, peppermint
MeSH Terms: conditions — Headache Disorders; Migraine Disorders; Headache | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- foot bath only (Placebo Comparator): 10 minute foot bath with addition of jojoba only
  Interventions: Other: foot bath
- foot bath and aromatherapy (Experimental): 10 minute foot bath with addition of jojoba with added Mentha piperita
  Interventions: Other: aromatherapy; Other: foot bath

INTERVENTIONS:
Other: aromatherapy
  Other Names: Mentha piperita
  Arms: foot bath and aromatherapy
Other: foot bath

SUMMARY:
The purpose of this study is to preliminarily establish the extent to which a brief aromatherapy intervention incrementally improves subjective and objective indicators of discomfort (pain, anxiety, and heart rate variability) beyond passive relaxation in youth with chronic headaches. A secondary objective is to establish the safety of using aromatherapy as a treatment strategy in youth with chronic headache. The investigators hypothesize that children randomized to the aromatherapy condition will demonstrate a greater improvement in pain, anxiety, and objectively measured distress (heart rate variability) than comparable children receiving only a passive relaxation treatment (a foot bath). The investigators further hypothesize that the aromatherapy intervention will be safe and well-tolerated by study participants.

DETAILED DESCRIPTION:
Complementary and alternative therapies play an increasing role in the multidisciplinary treatment of primary pediatric headache disorders. Every pediatric headache patient needs to have a personalized and tailored program of education, psychological strategies, pharmacotherapy and complementary medicine choices. This particular study may prove desirable for parents of children and adolescents with chronic headache. As documented by Termine, C., Ferrari, Ginevra, O., D'Arrigo, S., Rossi, M., & Lanzi, G. (2005), parents are often uncertain and fearful of submitting their children to treatment with traditional drugs, adolescents can use alternative therapies as a way of affirming their independence, and there are fewer drugs available to treat headache in children. Moreover, there is a 30-40% placebo response in headache sufferers (Mauskop, 2001). Children and adolescents should not be prevented from using alternative treatments, specifically essential oils, provided that the intervention is not harmful or costly. It is hoped this study will contribute to the scant research that exists and help define the indications, effects and limitations of aromatherapy use.

ELIGIBILITY:
Inclusion Criteria:

* • Male or female, children and adolescents age 7-17 years of age

  * Diagnosed with status migrainosus or refractory chronic daily headache according to the International Headache Society (ICHD-II) criteria. (A debilitating migraine lasting for more than 72 hours or a headache that lasts hours or may be continuous occurring on > 15 days per month for > 3 months.)
  * No prior history of aromatherapy / essential oil use
  * Able to read, comprehend and complete study procedures. Capable of reading and completing all subjective measures in English
  * Are sufficiently alert to be assessed and communicate
  * Must be compliant with routine medical care and able to perform study-related procedures
  * Provide written informed consent from parent/legal guardian and child assent in accordance with IRB regulations

Exclusion Criteria:

* • Known sensitivity to essential oils

  * History of cardiac fibrillation
  * History of G6PD deficiency
  * History of uncontrolled asthma (current, active wheezing)
  * History of diabetes, high blood pressure, epilepsy,
  * Inflammatory or sensory limitations of lower extremities or concurrent lesions of the foot(s)
  * Past or concurrent history of olfactory impairment
  * Concomitant use of propanolol
  * Tobacco use
  * Hepatotoxicity
  * Pregnancy

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2015-03-25 (Actual); Primary Completion 2017-01-04 (Actual); Study Completion 2017-01-04 (Actual)

PRIMARY OUTCOMES:
improvement in subjective and objective indicators of discomfort | 30 minutes
  pain and anxiety measured subjectively via VAS
improvement in subjective and objective indicators of discomfort | 30 minutes
  heart rate variability measured -10, 10 and 20 minutes

SECONDARY OUTCOMES:
number of Adverse Events | 30 minutes
  assessment of presence or absence of Adverse Events or Serious Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Rae A Kingsley, MSN, APRN, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Background] Battaiglia, S. (2003). The complete guide to aromatherapy (2nd edition). Brisbane, Australia: The International Centre of Holistic Aromatherapy
- [Background] Blume HK. Pediatric headache: a review. Pediatr Rev. 2012 Dec;33(12):562-76. doi: 10.1542/pir.33-12-562. No abstract available. PMID 23204398
- [Background] Buckle J. Use of aromatherapy as a complementary treatment for chronic pain. Altern Ther Health Med. 1999 Sep;5(5):42-51. PMID 10484830
- [Background] Fitzgerald M, Culbert T, Finkelstein M, Green M, Liu M. The effect of gender and ethnicity on children's attitudes and preferences for essential oils: a follow up study. Explore (NY). 2010 May-Jun;6(3):172. doi: 10.1016/j.explore.2010.02.002. No abstract available. PMID 20451151
- [Background] Gardiner P, Wornham W. Recent review of complementary and alternative medicine used by adolescents. Curr Opin Pediatr. 2000 Aug;12(4):298-302. doi: 10.1097/00008480-200008000-00002. PMID 10943807
- [Background] Gaul C, Eismann R, Schmidt T, May A, Leinisch E, Wieser T, Evers S, Henkel K, Franz G, Zierz S. Use of complementary and alternative medicine in patients suffering from primary headache disorders. Cephalalgia. 2009 Oct;29(10):1069-78. doi: 10.1111/j.1468-2982.2009.01841.x. Epub 2009 Apr 2. PMID 19366356
- [Background] Gobel H, Schmidt G, Soyka D. Effect of peppermint and eucalyptus oil preparations on neurophysiological and experimental algesimetric headache parameters. Cephalalgia. 1994 Jun;14(3):228-34; discussion 182. doi: 10.1046/j.1468-2982.1994.014003228.x. PMID 7954745
- [Background] Halcon LL. Aromatherapy: therapeutic applications of plant essential oils. Minn Med. 2002 Nov;85(11):42-6. PMID 12498066
- [Background] Kabbouche MA, Linder SL. Acute treatment of pediatric headache in the emergency department and inpatient settings. Pediatr Ann. 2005 Jun;34(6):466-71. doi: 10.3928/0090-4481-20050601-12. PMID 16018229
- [Background] Keifer D, Ulbricht C, Abrams TR, Basch E, Giese N, Giles M, DeFranco Kirkwood C, Miranda M, Woods J. Peppermint (Mentha piperita): an evidence-based systematic review by the Natural Standard Research Collaboration. J Herb Pharmacother. 2007;7(2):91-143. doi: 10.1300/j157v07n02_07. PMID 18285310
- [Background] Kligler B, Chaudhary S. Peppermint oil. Am Fam Physician. 2007 Apr 1;75(7):1027-30. PMID 17427617
- [Background] Lee MS, Choi J, Posadzki P, Ernst E. Aromatherapy for health care: an overview of systematic reviews. Maturitas. 2012 Mar;71(3):257-60. doi: 10.1016/j.maturitas.2011.12.018. Epub 2012 Jan 27. PMID 22285469
- [Background] Lewis D, Ashwal S, Hershey A, Hirtz D, Yonker M, Silberstein S; American Academy of Neurology Quality Standards Subcommittee; Practice Committee of the Child Neurology Society. Practice parameter: pharmacological treatment of migraine headache in children and adolescents [RETIRED]: report of the American Academy of Neurology Quality Standards Subcommittee and the Practice Committee of the Child Neurology Society. Neurology. 2004 Dec 28;63(12):2215-24. doi: 10.1212/01.wnl.0000147332.41993.90. PMID 15623677
- [Background] Loman DG. The use of complementary and alternative health care practices among children. J Pediatr Health Care. 2003 Mar-Apr;17(2):58-63. doi: 10.1067/mph.2003.29. PMID 12665727
- [Background] Martin, I. (2007). Aromatherapy for Massage Practitioners. Lippincott Williams Wilkins; Baltimore, MD.
- [Background] Mauskop A. Alternative therapies in headache. Is there a role? Med Clin North Am. 2001 Jul;85(4):1077-84. doi: 10.1016/s0025-7125(05)70360-6. PMID 11480259
- [Background] Mosby Skills Adapted from Perry, A.G., Potter, P.A., Ostendorf, W.R. (2014). Clinical nursing skills & techniques (8th ed.). St. Louis: Mosby
- [Background] Nishimura M, Tatsuya Saito TS, Kato T, Onodera S. Effects of Water Temperature during Foot Bath in Young Females. Yonago Acta Med. 2013 Sep;56(3):79-80. Epub 2013 Sep 11. PMID 24174706
- [Background] Peterson CC, Palermo TM. Parental reinforcement of recurrent pain: the moderating impact of child depression and anxiety on functional disability. J Pediatr Psychol. 2004 Jul-Aug;29(5):331-41. doi: 10.1093/jpepsy/jsh037. PMID 15187172
- [Background] Posadzki P, Alotaibi A, Ernst E. Adverse effects of aromatherapy: a systematic review of case reports and case series. Int J Risk Saf Med. 2012 Jan 1;24(3):147-61. doi: 10.3233/JRS-2012-0568. PMID 22936057
- [Background] Roth-Isigkeit A, Thyen U, Stoven H, Schwarzenberger J, Schmucker P. Pain among children and adolescents: restrictions in daily living and triggering factors. Pediatrics. 2005 Feb;115(2):e152-62. doi: 10.1542/peds.2004-0682. PMID 15687423
- [Background] Saeki Y. The effect of foot-bath with or without the essential oil of lavender on the autonomic nervous system: a randomized trial. Complement Ther Med. 2000 Mar;8(1):2-7. PMID 10812753
- [Background] Saeki Y, Nagai N, Hishinuma M. Effects of footbathing on autonomic nerve and immune function. Complement Ther Clin Pract. 2007 Aug;13(3):158-65. doi: 10.1016/j.ctcp.2006.12.006. Epub 2007 Feb 20. PMID 17631258
- [Background] Schetzek S, Heinen F, Kruse S, Borggraefe I, Bonfert M, Gaul C, Gottschling S, Ebinger F. Headache in children: update on complementary treatments. Neuropediatrics. 2013 Feb;44(1):25-33. doi: 10.1055/s-0032-1333435. Epub 2013 Jan 11. PMID 23315555
- [Background] Smith MC, Kyle L. Holistic foundations of aromatherapy for nursing. Holist Nurs Pract. 2008 Jan-Feb;22(1):3-9; quiz 10-1. doi: 10.1097/01.HNP.0000306321.03590.32. PMID 18172401
- [Background] Stankewitz A, May A. Increased limbic and brainstem activity during migraine attacks following olfactory stimulation. Neurology. 2011 Aug 2;77(5):476-82. doi: 10.1212/WNL.0b013e318227e4a8. Epub 2011 Jul 20. PMID 21775739
- [Background] Szema AM, Barnett T. Allergic reaction to mint leads to asthma. Allergy Rhinol (Providence). 2011 Jan;2(1):43-5. doi: 10.2500/ar.2011.2.0008. PMID 22852115
- [Background] Termine C, Ginevra OF, D'Arrigo S, Rossi M, Lanzi G. Alternative therapies in the treatment of headache in childhood, adolescence and adulthood. Funct Neurol. 2005 Jan-Mar;20(1):9-14. PMID 15948561
- [Background] Tisserand, R. & Balacs, T. (1995). Essential oil safety. Edinburgh: Churchill Livingstone
- [Background] Tisserand, R. & Young, R. (2014). Essential Oil Safety. A Guide for Health Care Professionals (2nd edition). Elsevier
- [Background] von Baeyer CL. Interpreting the high prevalence of pediatric chronic pain revealed in community surveys. Pain. 2011 Dec;152(12):2683-2684. doi: 10.1016/j.pain.2011.08.023. Epub 2011 Sep 14. No abstract available. PMID 21920669
- [Derived] Kingsley RA. Randomized Trial Examining Efficacy of Mentha piperita in Reducing Chronic Headache Discomfort in Youth. Pain Manag Nurs. 2023 Dec;24(6):e139-e147. doi: 10.1016/j.pmn.2023.08.004. Epub 2023 Sep 18. PMID 37730471
- See also: developing and delivering research-based, practical, and reliable tools and technologies — http://www.heartmath.com
- See also: headache classification — http://ihs-classification.org/en/
- See also: Aromatherapy and Essential Oils (PDQ). National Cancer Institute at the National Institutes of Health — http://www.cancer.gov/cancertopics/pdq/cam/aromatherapy/healthprofessional/
- See also: Peppermint oil (Mentha x piperita L.). Natural Standard Database Web site. — http://www.naturalstandard.com
- See also: Research Randomizer ©1997-2008 by Geoffery C. Urbaniak and Scott Plous Social Psychology Network — http://www.randomizer.org/